CLINICAL TRIAL: NCT04795492
Title: Effect of Remote Intervention in Patients With SCAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough patients
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Weihua Song, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERIP
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Stable Chronic Angina; Ischemic Heart Disease; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Angina, Stable; Myocardial Ischemia; Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Remote intervention
  Interventions: Behavioral: remote intervention
- Control group (Active Comparator): Routine outpatient follow-up
  Interventions: Behavioral: Routine outpatient follow-up

INTERVENTIONS:
Behavioral: remote intervention — Medication adherence and risk factor modification status were assessed, then individualized feedback, encouragement and recommendations were provided. Risk factor modification included lipid control, smoking and drinking cessation, BP monitoring, dietary change keeping a healthy weight and in our trial. There were also a lot of educational materials about coronary heart disease knowledge that were reviewed by cardiologists, and participants were free to provide them whenever and wherever they want.
  Arms: Intervention group
Behavioral: Routine outpatient follow-up — Participants in this group received standard outpatient cardiology follow-up with formal cardiac rehabilitation and secondary prevention.
  Arms: Control group

SUMMARY:
The study was a multicenter, two-arm, parallel, open-label, prospective clinical trial that evaluated a remote intervention with 1 year of follow-up.

DETAILED DESCRIPTION:
Objective: This study is intended to verify the effect of a remote intervention on adherence to drugs and risk factors control in patients with stable coronary artery disease.

Study design: The study was a multicenter, two-arm, parallel, open-label, prospective clinical trial that evaluated the effect of a remote intervention on adherence to drugs and risk factors control in patients with stable coronary artery disease with 1 year of follow-up.

Study intervention: Participants in the experimental group received remote guidance from the cardiac rehabilitation team in the community hospital every month after enrollment. The control group had no special intervention. All patients received follow-up at 6 months and 1-year follow-up.

Outcome measures: The primary outcome was medication adherence. Secondary outcomes included smoking, drinking, blood pressure, body mass index, LDL cholesterol, HbA1c, and major adverse cerebral cardiovascular events(MACCE). Medication compliance consists of the following five medications: aspirin, P2Y12 receptor antagonist, statin, ACEI/ARB and beta-blocker.

Statistical analysis: Values of analyzed endpoints between intervention group and control group will be compared according to the analysis plan. We'll follow a prespecified analysis plan and subgroup analysis will be conducted accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-99 years
2. Diagnosed with SCAD according to guidelines by coronary CTA or coronary angiography (including stable angina, ischemic cardiomyopathy, and the stable course after acute coronary syndrome)
3. Have sufficient Chinese language proficiency to reading, speaking and listening
4. Live with at least one caregiver or guardian in the household
5. Presence of stable hemodynamics without using vasopressor
6. Able to individually consent
7. Not participating in any other clinical trial

Exclusion Criteria:

1. Unable to provide informed consent
2. Unable to be involved in clinical follow-up and treatment
3. Suffered comorbidity with a life expectancy of less than 1 year
4. Have contra-indication to cardiac rehabilitation
5. Acute coronary syndrome
6. History of noncompliance with medical therapy
7. Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial
8. Planned major surgery necessitating interruption of antiplatelet therapy
9. Inability to comply with the protocol
10. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest of the subject or that could prevent, limit or confound the protocol-specified assessments

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 1 year
  Compliance and administration of cardiovascular protective drugs

SECONDARY OUTCOMES:
Blood Pressure | 1 year
  BP was measured twice by an electronic device after 10 min of seated rest and calculated as the mean of 2 measurements
Body Mass Index | 1 year
  standard protocol
LDL Cholesterol | 1 year
  standard protocol
HbA1c | 1 year
  standard protocol
Smoking | 1 year
  self-reported
Drinking | 1 year
  self-reported
Aspirin | 1 year
  self-reported
P2Y12 receptor antagonist | 1 year
  self-reported
Statin | 1 year
  self-reported
ACEI/ARB | 1 year
  self-reported
Beta-blocker | 1 year
  self-reported
MACCE | 1 year
  acute myocardial infarction, acute heart failure, rehospitalization for cardiovascular event, stroke, death from any cause, death from a cardiovascular cause and unplanned revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Song, MD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Science; National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Science; National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng X, Spatz ES, Bai X, Huo X, Ding Q, Horak P, Wu X, Guan W, Chow CK, Yan X, Sun Y, Wang X, Zhang H, Liu J, Li J, Li X, Spertus JA, Masoudi FA, Krumholz HM. Effect of Text Messaging on Risk Factor Management in Patients With Coronary Heart Disease: The CHAT Randomized Clinical Trial. Circ Cardiovasc Qual Outcomes. 2019 Apr;12(4):e005616. doi: 10.1161/CIRCOUTCOMES.119.005616. PMID 30998400
- [Background] Yu C, Liu C, Du J, Liu H, Zhang H, Zhao Y, Yang L, Li X, Li J, Wang J, Wang H, Liu Z, Rao C, Zheng Z; MISSION-2 Collaborative Group. Smartphone-based application to improve medication adherence in patients after surgical coronary revascularization. Am Heart J. 2020 Oct;228:17-26. doi: 10.1016/j.ahj.2020.06.019. Epub 2020 Jul 4. PMID 32745732
- [Background] Chen X, Zhou X, Li H, Li J, Jiang H. The value of WeChat application in chronic diseases management in China. Comput Methods Programs Biomed. 2020 Nov;196:105710. doi: 10.1016/j.cmpb.2020.105710. Epub 2020 Aug 14. PMID 32858284